CLINICAL TRIAL: NCT04557098
Title: A Phase 1/2, First-in-Human, Open-Label, Dose Escalation Study of Teclistamab, a Humanized BCMA x CD3 Bispecific Antibody, in Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Teclistamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MajesTEC-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108859; TECLIMMY1001-P3 (Other: Janssen Research & Development, LLC); 2016-002122-36 (EudraCT Number); 2023-503438-40-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-09-17; First posted 2020-09-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 3: Teclistamab (Experimental): Participants will receive teclistamab subcutaneously (SC) at recommended Phase 2 dose (RP2D) in Cohort A and Cohort C.
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered SC.
  Other Names: JNJ-64007957

SUMMARY:
The purpose of this study is to evaluate the efficacy of teclistamab at the recommended Phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria: -

* Documented diagnosis of multiple myeloma according to IMWG diagnostic criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Measurable disease: Cohort A and Cohort C: Multiple myeloma must be measurable by central laboratory assessment
* A female participant of childbearing potential must have a negative pregnancy test at screening
* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Cohort A: received at least >=3 prior lines of therapy and previously received a PI, an IMiD and an anti-CD38 monoclonal antibody; Cohort C: received >= 3 prior lines of therapy that included a PI, an IMiD, an anti-CD38 monoclonal antibody, and an anti-B cell maturation antigen (BCMA) treatment (with CART-T cells or an antibody drug conjugate (ADC)

Exclusion Criteria:

* Plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome, or primary amyloid light-chain amyloidosis
* The following medical conditions: Pulmonary compromise requiring supplemental oxygen use to maintain adequate oxygenation, human immunodeficiency virus (HIV) infection, hepatitis B or C infection, stroke or seizure less than or equal to (<=) 6 m, autoimmune disease, uncontrolled systemic infection, cardiac conditions (Myocardial Infarction <= 6 m, stage III-IV congestive heart failure, etc)
* Received any therapy that is targeted to BCMA, with the exception of Cohort C in Part 3
* Prior antitumor therapy, within 21 days (PI or radiotherapy within 14 days, IMiDs within 7 days, Gene modified adoptive cell therapy within 3 months) prior to first dose of study drug
* Toxicities from previous anticancer therapies that have not resolved to baseline or to <= grade 1 (except for alopecia or peripheral neuropathy)
* Received a cumulative dose of corticosteroids equivalent to >=140 mg of prednisone within the 14-day period before the first dose of study drug (does not include pretreatment medication)
* Known active central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma (MM)
* Myelodysplastic syndrome or active malignancies other than relapsed/refractory multiple myeloma with exceptions are: 1) Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured 2) Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured. 3) Noninvasive cervical cancer treated within the last 24 months that is considered completely cured. 4) Localized prostate cancer (N0M0) 5) Breast cancer: Adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence. 6) Malignancy that is considered cured with minimal risk of recurrence
* Prior allogenic stem cell transplant <=6 months
* Prior autologous stem cell transplant <=12 weeks
* Live, attenuated vaccine within 4 weeks prior to the first dose of teclistamab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2027-05-28 (Estimated)

PRIMARY OUTCOMES:
Cohorts A and C: Overall Response Rate (ORR) | Up to 2.9 years
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Cohorts A and C: Duration of Response (DOR) | Up to 2.9 years
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria, or death due to PD, whichever occurs first.
Cohorts A and C: Very Good Partial Response (VGPR) or Better Rate | Up to 2.9 years
  VGPR or better rate is defined as the percentage of patients who achieve a VGPR or better according to IMWG response criteria.
Cohorts A and C: Cohorts A and C: Complete Response (CR) or Better Rate | Up to 2.9 years
  CR or better rate is defined as the percentage of patients who achieve a complete response (CR) or better according to IMWG response criteria.
Cohorts A and C: Stringent Complete Response (sCR) Rate | Up to 2.9 years
  sCR rate is defined as the percentage of patients who achieve a stringent complete response (sCR) according to IMWG response criteria.
Cohorts A and C: Time to Response (TTR) | Up to 2.9 years
  TTR is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.
Cohorts A and C: Progression-free Survival (PFS) | Up to 2.9 years
  PFS is defined as the time from the date of first dose of study drug to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Cohorts A and C: Overall Survival (OS) | Up to 2.9 years
  OS is defined as the time from the date of first dose of study drug to the date of the participant's death.
Cohorts A and C: Minimal Residual Disease (MRD) Negative Rate | Up to 2.9 years
  MRD-negative rate is defined as the proportion of participants who achieved MRD-negative status to a threshold of 10^-5 at any timepoint after initial dose of teclistamab and before disease progression or starting subsequent therapy
Cohorts A and C: Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 2.9 years
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Cohorts A and C: Number of Participants with Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability | Up to 2.9 years
  An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Cohorts A and C: Number of Participants with AEs by Severity | Up to 2.9 years
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Cohorts A and C: Number of Participants with Laboratory Abnormalities in Clinical Laboratory Values | Up to 2.9 years
  Number of participants with laboratory abnormalities in clinical laboratory values (such as hemoglobin, platelets) will be reported.
Cohorts A and C: Serum Concentration of Teclistamab | Up to 3 months
  Serum concentrations of teclistamab will be reported.
Cohorts A and C: Number of Participants with Teclistamab Antibodies | Up to 2.9 years
  Antibodies to teclistamab will be assessed to evaluate potential immunogenicity.
Cohorts A and C: Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 item (EORTC QLQ-C30) | Baseline, up to 2.9 years
  The EORTC- QLQ-Core-30 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The recall period is 1 week ("past week"), and responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Cohorts A and C: Change from Baseline in HRQoL as Assessed by EuroQol Five Dimension Five Level Questionnaire (EQ-5D-5L) | Baseline, up to 2.9 years
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The scores for the 5 separate questions are categorical and cannot be analyzed as cardinal numbers.
Cohorts A and C: Change from Baseline in HRQoL as Assessed by Patient Global Impression of Severity (PGIS) | Baseline, up to 2.9 years
  The PGIS is a single item that assesses severity of the participant's health state, on a 5-point verbal rating scale. Score ranges from 1 (None) to 5 (Very Severe).
Cohorts A and C: Overall Response Rate (ORR) in Participants with High-risk Molecular Features | Up to 2.9 years
  ORR in participants with high risk is defined as the overall response rate among the high-risk molecular subgroups (del17p, t(4;14), t(14;16), or other high-risk molecular subtypes).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (51):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai Program for the Protection of Human Subjects, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Belgium (2):
  - Universitair Ziekenhuis Gent - UZ GENT, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network UHN Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (8):
  - Peking University First Hospital, Beijing
  - West China Hospital Si Chuan University, Chengdu
  - Sun Yat -Sen University Cancer Center, Guangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Shanghai Changzheng Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- France (6):
  - Centre Hospitalier Régional Universitaire de Lille, Hôpital Claude Huriez, Lille
  - Centre Hospitalier Lyon Sud, Lyon
  - C.H.U. Hotel Dieu - France, Nantes
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - Pôle IUC Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau, Tours
- Germany (4):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia Seràgnoli azienda ospedaliera univeristaria Policlinico S.Orsola-Malpighi, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
- VU Medisch Centrum, Amsterdam, Netherlands
- Spain (7):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Skane University Hospital, Lund
  - Haematology Centre, R 51, Stockholm
- United Kingdom (3):
  - University College Hospital, London
  - University Hospital Southampton, Sothampton
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinicaltrials/ transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Martin TG, van de Donk NWCJ, Rodriguez-Otero P, Mateos MV, Kobos R, Chastain K, Doyle M, Nooka AK. Plain language summary of the management of certain side effects of teclistamab in people with multiple myeloma. Future Oncol. 2026 Jan 23:1-13. doi: 10.1080/14796694.2025.2597732. Online ahead of print. PMID 41574880
- [Derived] Martin TG, Mateos MV, Yi JH, van de Donk NWCJ, Cai Z, Fu W, Garfall AL, Iida S, Jung SH, Kuroda Y, Niu T, Nooka AK, Min CK, Sidana S, Chastain K, Doyle M, Nishikawa K, Wang X, Song Y, Yamazaki H, Izumi Y, Zhuo J, Zhu A, Yoon DH, Du J, Ishida T. Efficacy and safety of teclistamab in triple-class exposed relapsed/refractory multiple myeloma: Pooled findings from three clinical cohorts and a retrospective cohort. Cancer. 2026 Jan 1;132(1):e70237. doi: 10.1002/cncr.70237. PMID 41485109
- [Derived] Gordan LN, Bensimon AG, Mu F, Kim N, Wu B, Lin D, Paner A, Fowler J, Marshall A, Van Sanden S, Ammann E, Goble J, Zhang X, Le HH, Min EE, Garrison LP Jr. Cost per responder for teclistamab and elranatamab in relapsed or refractory multiple myeloma in the United States. J Med Econ. 2025 Dec;28(1):910-920. doi: 10.1080/13696998.2025.2514909. Epub 2025 Jun 14. PMID 40495704
- [Derived] Guo Y, Niu J, Carde NAQ, Wu L, Miao X, Hanson S, Su Y, Ruixo CP, Vishwamitra D, Chastain K, Samtani MN, Wang W, Haddish-Berhane N. Teclistamab Dosing in Responders: Modeling and Simulation Results from the MajesTEC-1 Study in Relapsed/Refractory Multiple Myeloma. Target Oncol. 2025 Jul;20(4):651-661. doi: 10.1007/s11523-025-01149-1. Epub 2025 May 7. PMID 40332715
- [Derived] Touzeau C, Krishnan AY, Moreau P, Perrot A, Usmani SZ, Manier S, Cavo M, Martinez Chamorro C, Nooka AK, Martin TG, Karlin L, Leleu X, Bahlis NJ, Besemer B, Pei L, Stein S, Wang Lin SX, Trancucci D, Verona RI, Girgis S, Miao X, Uhlar CM, Chastain K, Garfall AL. Efficacy and safety of teclistamab in patients with relapsed/refractory multiple myeloma after BCMA-targeting therapies. Blood. 2024 Dec 5;144(23):2375-2388. doi: 10.1182/blood.2023023616. PMID 39172760
- [Derived] Cortes-Selva D, Perova T, Skerget S, Vishwamitra D, Stein S, Boominathan R, Lau O, Calara-Nielsen K, Davis C, Patel J, Banerjee A, Stephenson T, Uhlar C, Kobos R, Goldberg J, Pei L, Trancucci D, Girgis S, Wang Lin SX, Wu LS, Moreau P, Usmani SZ, Bahlis NJ, van de Donk NWCJ, Verona RI. Correlation of immune fitness with response to teclistamab in relapsed/refractory multiple myeloma in the MajesTEC-1 study. Blood. 2024 Aug 8;144(6):615-628. doi: 10.1182/blood.2023022823. PMID 38657201
- [Derived] Moreau P, Mateos MV, Gonzalez Garcia ME, Einsele H, De Stefano V, Karlin L, Lindsey-Hill J, Besemer B, Vincent L, Kirkpatrick S, Delforge M, Perrot A, van de Donk NWCJ, Pawlyn C, Manier S, Leleu X, Martinez-Lopez J, Ghilotti F, Diels J, Morano R, Albrecht C, Strulev V, Haddad I, Pei L, Kobos R, Smit J, Slavcev M, Marshall A, Weisel K. Comparative Effectiveness of Teclistamab Versus Real-World Physician's Choice of Therapy in LocoMMotion and MoMMent in Triple-Class Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Feb;41(2):696-715. doi: 10.1007/s12325-023-02738-0. Epub 2023 Dec 19. PMID 38110653
- [Derived] Martin TG, Moreau P, Usmani SZ, Garfall A, Mateos MV, San-Miguel JF, Oriol A, Nooka AK, Rosinol L, Chari A, Karlin L, Krishnan A, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Delforge M, Trancucci D, Pei L, Kobos R, Fastenau J, Gries KS, van de Donk NWCJ. Teclistamab Improves Patient-Reported Symptoms and Health-Related Quality of Life in Relapsed or Refractory Multiple Myeloma: Results From the Phase II MajesTEC-1 Study. Clin Lymphoma Myeloma Leuk. 2024 Mar;24(3):194-202. doi: 10.1016/j.clml.2023.11.001. Epub 2023 Nov 14. PMID 38052709
- [Derived] Frerichs KA, Verkleij CPM, Mateos MV, Martin TG, Rodriguez C, Nooka A, Banerjee A, Chastain K, Perales-Puchalt A, Stephenson T, Uhlar C, Kobos R, van der Holt B, Kruyswijk S, Kuipers MT, Groen K, Vishwamitra D, Skerget S, Cortes-Selva D, Doyle M, Zaaijer HL, Zweegman S, Verona RI, van de Donk NWCJ. Teclistamab impairs humoral immunity in patients with heavily pretreated myeloma: importance of immunoglobulin supplementation. Blood Adv. 2024 Jan 9;8(1):194-206. doi: 10.1182/bloodadvances.2023011658. PMID 38052042
- [Derived] Nooka AK, Rodriguez C, Mateos MV, Manier S, Chastain K, Banerjee A, Kobos R, Qi K, Verona R, Doyle M, Martin TG, van de Donk NWCJ. Incidence, timing, and management of infections in patients receiving teclistamab for the treatment of relapsed/refractory multiple myeloma in the MajesTEC-1 study. Cancer. 2024 Mar 15;130(6):886-900. doi: 10.1002/cncr.35107. Epub 2023 Nov 14. PMID 37960969
- [Derived] Miao X, Wu LS, Lin SXW, Xu Y, Chen Y, Iwaki Y, Kobos R, Stephenson T, Kemmerer K, Uhlar CM, Banerjee A, Goldberg JD, Trancucci D, Apte A, Verona R, Pei L, Desai R, Hickey K, Su Y, Ouellet D, Samtani MN, Guo Y, Garfall AL, Krishnan A, Usmani SZ, Zhou H, Girgis S. Population Pharmacokinetics and Exposure-Response with Teclistamab in Patients With Relapsed/Refractory Multiple Myeloma: Results From MajesTEC-1. Target Oncol. 2023 Sep;18(5):667-684. doi: 10.1007/s11523-023-00989-z. Epub 2023 Sep 15. PMID 37713090
- [Derived] Moreau P, van de Donk NW, Nahi H, Oriol A, Nooka AK, Martin T, Rosinol L, Karlin L, Benboubker L, Mateos MV, Popat R, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Olyslager Y, Uhlar C, Stephenson T, Rampelbergh RV, Banerjee A, Kobos R, Usmani SZ. Plain language summary of the MajesTEC-1 study of teclistamab for the treatment of people with relapsed or refractory multiple myeloma. Future Oncol. 2023 Apr;19(12):811-818. doi: 10.2217/fon-2023-0171. Epub 2023 May 3. PMID 37132225
- [Derived] Martin TG, Mateos MV, Nooka A, Banerjee A, Kobos R, Pei L, Qi M, Verona R, Doyle M, Smit J, Sun W, Trancucci D, Uhlar C, van de Donk NWCJ, Rodriguez C. Detailed overview of incidence and management of cytokine release syndrome observed with teclistamab in the MajesTEC-1 study of patients with relapsed/refractory multiple myeloma. Cancer. 2023 Jul 1;129(13):2035-2046. doi: 10.1002/cncr.34756. Epub 2023 Mar 29. PMID 36991547
- [Derived] Moreau P, van de Donk NWCJ, Delforge M, Einsele H, De Stefano V, Perrot A, Besemer B, Pawlyn C, Karlin L, Manier S, Leleu X, Weisel K, Ghilotti F, Diels J, Elsada A, Morano R, Strulev V, Pei L, Kobos R, Smit J, Slavcev M, Mateos MV. Comparative Efficacy of Teclistamab Versus Current Treatments in Real-World Clinical Practice in the Prospective LocoMMotion Study in Patients with Triple-Class-Exposed Relapsed and/or Refractory Multiple Myeloma. Adv Ther. 2023 May;40(5):2412-2425. doi: 10.1007/s12325-023-02480-7. Epub 2023 Mar 24. PMID 36961654
- [Derived] Moreau P, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Nooka AK, Martin T, Rosinol L, Chari A, Karlin L, Benboubker L, Mateos MV, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Verona R, Girgis S, Lin SXW, Olyslager Y, Jaffe M, Uhlar C, Stephenson T, Van Rampelbergh R, Banerjee A, Goldberg JD, Kobos R, Krishnan A, Usmani SZ. Teclistamab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2022 Aug 11;387(6):495-505. doi: 10.1056/NEJMoa2203478. Epub 2022 Jun 5. PMID 35661166
- See also: Dose Escalation Study of JNJ-64007957, a Humanized BCMA CD3 DuoBody® Antibody, in Participants With Relapsed or Refractory Multiple Myeloma — https://clinicaltrials.gov/ct2/show/NCT03145181